CLINICAL TRIAL: NCT05692154
Title: A Phase IIIb, Single-center, Double-blind, Two-arms, Placebo-controlled, Randomized, Parallel-group Clinical Trial to Evaluate the Efficacy and Safety of 2-day Pre-treatment With Fexofenadine in Patients Suffering From Seasonal Allergic Rhinitis
Brief Title: A Placebo-controlled Study of 2-day Pre-treatment With Fexofenadine in Seasonal Allergic Rhinitis
Acronym: FEXPRESAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Opella Healthcare Group SAS, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LPS17180; U1111-1278-3949 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — fexofenadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A (active-active) (Experimental): Two days of pre-treatment with Fexofenadine 180 mg each day in the morning on Day 2 and Day 3, then Fexofenadine180 mg after the pollen challenge on Day 4.
  Interventions: Drug: Fexofenadine
- Arm B (placebo-active) (Experimental): Two days of pre-treatment with tablet of matching placebo each day in the morning on Day 2 and Day 3, then Fexofenadine180 mg after the pollen challenge on Day 4.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fexofenadine — Fexofenadine oral tablet
  Arms: Arm A (active-active)
Drug: Placebo — Fexofenadine matching placebo oral tablet
  Arms: Arm B (placebo-active)

SUMMARY:
This study is a proof-of-concept study to demonstrate if a daily dose of a 2-days pre-treatment of Fexofenadine 180mg is effective in alleviating the AR symptoms and to assess the additional benefit to the patient in terms of preventing Allergic Rhinitis (AR) symptoms.

The total study duration per participant is expected at least 4 months, depending on the timing of the screening visit. 5 visits are planned, screening, confirmation inclusion challenge, randomization visit, challenge and end of study visit.

DETAILED DESCRIPTION:
The end of the study is defined as the date of the last visit of the last participant in the study.

A participant is considered to have completed the study if he/she has completed all visits of the study including Visit 5 (Day 5).

ELIGIBILITY:
Inclusion Criteria:

* Participants are eligible to be included in the study only if all of the following criteria apply:
* Participant is willing to provide written informed consent.
* Adult participants (18 to 80 years old) suffering from seasonal allergic rhinitis (SAR) provoked by Ragweed pollen.
* Participants having a total nasal symptom score (TNSS)-3 ≥4 (with 3 nasal symptoms) at first pollen challenge at Visit 2.
* Having a 2-year history of SAR with Positive skin prick test to Ragweed allergen at screening (with a wheal diameter at least 3 mm larger than that produced by the negative control).

Exclusion Criteria:

* History of anaphylaxis to Ragweed pollen History of asthma or exacerbations in the past 12 months requiring regular inhaled corticosteroids for greater than 4 weeks per year, any oral corticosteroid usage, any emergency department visit for asthma or any asthma-related hospitalization. Mild asthmatics treated only with pro re nata short-acting β2agonists, less than 2 doses per week can be enrolled.
* History of chronic sinusitis, defined as a sinus symptoms lasting greater than 12 weeks that includes 2 or more major factors or 1 major factor and 2 minor factors. Major factors are defined as facial pain or pressure, nasal obstruction or blockage, nasal discharge or purulence or discolored postnasal discharge, purulence in nasal cavity, or impaired or loss of smell. Minor factors are defined as headache, fever, halitosis, fatigue, dental pain, cough, and ear pain, pressure, or fullness.
* History of systemic disease affecting the immune system such as autoimmune diseases, immune complex disease, or immunodeficiency, where, in the opinion of the study physician, participation in the trial would pose a risk or significant effect on the immune system.
* Presence or history of drug hypersensitivity to fexofenadine and/or its excipients.
* Participants unable to stop the following forbidden treatments/nutriments prior to pollen challenge:

  * Antihistamines: within 3 days for first-generation antihistamines, within 2 days for second-generation antihistamines.
  * Intranasal or inhaled corticosteroids: 7 days.
  * Ocular, intranasal, or inhaled sodium cromoglycate: 14 days.
  * High doses of systemic corticosteroids: 30 days.
  * Leukotriene antagonists: 30 days.
  * Intranasal or systemic decongestants: 3 days.
  * Tricyclic antidepressants: 7 days.
  * Any citrus fruits (grapefruit, orange, etc.) or their juices, as well as all fruit juices: 5 days.
  * Aluminum-and-magnesium containing antacids: 7 days.
  * Omalizumab/dupilumab: within 6 months
* Any contraindications to fexofenadine, according to the labeling.
* The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2023-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number : 1240001, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: LPS17180 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25295&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 95 participants took part in the study at one investigative site in Canada from 23 January 2023 to 14 March 2023.
Pre-assignment Details: Participants suffering from seasonal allergic rhinitis were randomly assigned in a 1:1 ratio to two arm groups Fexofenadine Pre-Treatment and Placebo Pre-Treatment.
Period: Overall Study
Arm/Group | Arm A (Active-active) | Arm B (Placebo-active)
Started | 47 | 48
Intent To Treat (ITT) Analysis Set (The ITT set contained all eligible participants (passed screening and confirmation challenge) who had been allocated to a randomized treatment regardless of whether study drug wallet was used or not.) | 47 | 48
Safety Analysis (SAF) Set (The SAF set contained all participants in the ITT set who received at least one dose of study drug and participants were classified according to treatment received.) | 47 | 47 (One participant did not receive study treatment and had been excluded from SAF.)
Modified Intent-to-Treat (mITT) Analysis Set (The mITT analysis set contained all eligible, ITT, and treated participants with Total Nasal Symptom Score of 3 symptoms (TNSS-3) evaluation Hour 0 (H0) at visit 4 (V4) and at least a further time point at Visit 4.) | 47 | 47
Completed | 47 | 47
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: The mITT analysis set contained all eligible, ITT, and treated participants with Total Nasal Symptom Score of 3 symptoms (TNSS-3) evaluation Hour 0 (H0) at visit 4 (V4) and at least a further time point at Visit 4.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Active-active) | Arm B (Placebo-active) | Total
Number analyzed (Participants) | 47 | 47 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.0 (12.82) | 44.7 (13.05) | 45.9 (12.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 34 | 68
  Male | 13 | 13 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 47 | 46 | 93
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 41 | 45 | 86
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Area Under Curve (AUC) of the Total Nasal Symptoms Score (TNSS-3)
Description: TNSS-3=composite score calculated as sum of rhinorrhea, sneezing, and nasal itching scores (TNSS-3: scale of each symptom is scored from 0 to 3), where 0 indicates no symptoms, a score of 1 for mild symptoms that are easily tolerated, 2 for awareness of symptoms which are bothersome but tolerable and 3 is reserved for severe symptoms that are hard to tolerate and interfere with daily activity. Individual scores were collected in e-diary. AUC of TNSS from time of the first observation to time of the last observation (AUC [0-6 hr]) was calculated by using the linear trapezoid method. Trapezoidal rule involves dividing the area into a number of strips of equal width. Then, approximating the area of each strip by the area of the trapezium formed when a chord replaces upper end. Sum of these approximations gives final numerical result of area under the curve. AUC range: Arm A=0.0-43.5; Arm B=2.1-39.9.
Time Frame: From 0 hour to 6 hours at Day 4
Population: The mITT analysis set contained all eligible, ITT, and treated participants with TNSS-3 evaluation at H0 at V4 and at least a further time point at Visit 4.
Measure: Mean (Standard Deviation); unit: Sum of scores*hours
Arm/Group | Arm A (Active-active) | Arm B (Placebo-active)
Number analyzed (Participants) | 47 | 47
Sum of scores*hours | 16.96 (9.090) | 21.42 (10.431)
Statistical Analysis 1: Comparison: Arm A (Active-active) vs Arm B (Placebo-active); Test type: Superiority; p = 0.038, ANCOVA; Least Square Mean Difference = -4.24, 95% CI 2-sided [-8.24 to -0.23], Standard Error of Mean 2.015 — Least-squares means, standard errors and p-value are taken from an analysis of covariance model, with treatment group as fixed effect and baseline TNSS (H0 at Visit 4) as covariate

2. Secondary Outcome: AUC of Total Ocular Symptoms Score (TOSS) (H0-H6 at Day 4)
Description: TOSS=composite score calculated as the sum of red/burning eyes, tearing, itchy/watery eyes scores (TOSS: scale of each symptom is scored from 0 to 3), where 0 indicates no symptoms, a score of 1 for mild symptoms that are easily tolerated, 2 for awareness of symptoms which are bothersome but tolerable and 3 is reserved for severe symptoms that are hard to tolerate and interfere with daily activity. individual scores were collected in e-diary. AUC of TOSS from time of the first observation to time of the last observation (AUC [0-6 hr]) was calculated by using the linear trapezoid. Trapezoidal rule involves dividing the area into a number of strips of equal width. Then, approximating the area of each strip by the area of the trapezium formed when a chord replaces upper end. Sum of these approximations gives final numerical result of area under the curve. AUC range: Arm A=0.0-43.6; Arm B=0.0-35.1.
Time Frame: From 0 hour to 6 hours at Day 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Sum of scores*hours
Arm/Group | Arm A (Active-active) | Arm B (Placebo-active)
Number analyzed (Participants) | 47 | 47
Sum of scores*hours | 11.74 (10.451) | 16.21 (11.253)
Statistical Analysis 1: Comparison: Arm A (Active-active) vs Arm B (Placebo-active); Test type: Superiority; p = 0.025, ANCOVA; Least Square Mean Difference = -4.75, 95% CI 2-sided [-8.90 to -0.60], Standard Error of Mean 2.088 — Least-squares means, standard errors and p-value are taken from an analysis of covariance, with treatment group as fixed categorical effect and baseline TOSS (H0 at Visit 4) as covariate

3. Secondary Outcome: AUC of Total Nasal Symptoms Score (TNSS-3) (H0-H12 at Day 4)
Description: TNSS-3=composite score calculated as sum of rhinorrhea, sneezing, and nasal itching scores (TNSS-3: scale of each symptom is scored from 0 to 3), where 0 indicates no symptoms, a score of 1 for mild symptoms that are easily tolerated, 2 for awareness of symptoms which are bothersome but tolerable and 3 is reserved for severe symptoms that are hard to tolerate and interfere with daily activity. Individual scores were collected in e-diary. AUC of TNSS from time of the first observation to time of the last observation (AUC [0-12 hr]) was calculated by using the linear trapezoid method. Trapezoidal rule involves dividing the area into a number of strips of equal width. Then, approximating the area of each strip by the area of the trapezium formed when a chord replaces upper end. Sum of these approximations gives final numerical result of area under the curve. AUC range: Arm A=0.0-63.5; Arm B=2.1-69.4.
Time Frame: From 0 hour to 12 hours at Day 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Sum of scores*hours
Arm/Group | Arm A (Active-active) | Arm B (Placebo-active)
Number analyzed (Participants) | 47 | 47
Sum of scores*hours | 23.66 (14.049) | 31.01 (18.555)
Statistical Analysis 1: Comparison: Arm A (Active-active) vs Arm B (Placebo-active); Test type: Superiority; p = 0.048, ANCOVA; Least Square Mean Difference = -6.50, 95% CI 2-sided [-12.95 to -0.05], Standard Error of Mean 3.247 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: AUC of Total Ocular Symptoms Score (TOSS) (H0-H12 at Day 4)
Description: TOSS=composite score calculated as the sum of red/burning eyes, tearing, itchy/watery eyes scores (TOSS: scale of each symptom is scored from 0 to 3), where 0 indicates no symptoms, a score of 1 for mild symptoms that are easily tolerated, 2 for awareness of symptoms which are bothersome but tolerable and 3 is reserved for severe symptoms that are hard to tolerate and interfere with daily activity. individual scores were collected in e-diary. AUC of TOSS from time of the first observation to time of the last observation (AUC [0-12 hr]) was calculated by using the linear trapezoid. Trapezoidal rule involves dividing the area into a number of strips of equal width. Then, approximating the area of each strip by the area of the trapezium formed when a chord replaces upper end. Sum of these approximations gives final numerical result of area under the curve. AUC range: Arm A=0.0-58.6; Arm B=0.0-65.5.
Time Frame: From 0 hour to 12 hours at Day 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Sum of scores*hours
Arm/Group | Arm A (Active-active) | Arm B (Placebo-active)
Number analyzed (Participants) | 47 | 47
Sum of scores*hours | 14.74 (14.432) | 21.67 (17.154)
Statistical Analysis 1: Comparison: Arm A (Active-active) vs Arm B (Placebo-active); Test type: Superiority; p = 0.011, ANCOVA; Least Square Mean Difference = -7.47, 95% CI 2-sided [-13.21 to -1.73], Standard Error of Mean 2.890 — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: AUC of Total Nasal Symptoms Score (TNSS-3) (Day 1 to Day 4)
Description: TNSS-3=composite score calculated as sum of rhinorrhea, sneezing, and nasal itching scores (TNSS-3:scale of each symptom is scored from 0 to 3), where 0 indicates no symptoms, a score of 1 for mild symptoms that are easily tolerated, 2 for awareness of symptoms which are bothersome but tolerable and 3 is reserved for severe symptoms that are hard to tolerate and interfere with daily activity. Individual scores were collected in e-diary. AUC of TNSS from time of the first observation to time of the last observation (AUC [Day 1 to Day 4]) was calculated by using the linear trapezoid method. Trapezoidal rule involves dividing the area into a number of strips of equal width. Then, approximating the area of each strip by the area of the trapezium formed when a chord replaces upper end. Sum of these approximations gives final numerical result of area under the curve. AUC range: Arm A=0.0-267.8; Arm B=2.1-379.0.
Time Frame: From randomization (Day 1) to Day 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Sum of scores*hours
Arm/Group | Arm A (Active-active) | Arm B (Placebo-active)
Number analyzed (Participants) | 47 | 47
Sum of scores*hours | 56.34 (55.697) | 65.48 (76.454)
Statistical Analysis 1: Comparison: Arm A (Active-active) vs Arm B (Placebo-active); Test type: Superiority; p = 0.074, ANCOVA; Least Square Mean Difference = -18.45, 95% CI 2-sided [-38.74 to 1.83], Standard Error of Mean 10.211 — Least-squares means, standard errors and p-value are taken from an analysis of covariance, with treatment group as fixed categorical effect and baseline TNSS (Day 1) as covariate

6. Secondary Outcome: AUC of Total Ocular Symptoms Score (TOSS) (Day 1 to Day 4)
Description: TOSS=composite score calculated as the sum of red/burning eyes, tearing, itchy/watery eyes scores (TOSS: scale of each symptom is scored from 0 to 3), where 0 indicates no symptoms, a score of 1 for mild symptoms that are easily tolerated, 2 for awareness of symptoms which are bothersome but tolerable and 3 is reserved for severe symptoms that are hard to tolerate and interfere with daily activity. individual scores were collected in e-diary. AUC of TOSS from time of the first observation to time of the last observation (AUC [Day 1 to Day 4]) was calculated by using the linear trapezoid. Trapezoidal rule involves dividing the area into a number of strips of equal width. Then, approximating the area of each strip by the area of the trapezium formed when a chord replaces upper end. Sum of these approximations gives final numerical result of area under the curve. AUC range: Arm A=0.0-226.6; Arm B=0.0-304.5.
Time Frame: From randomization (Day 1) to Day 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Sum of scores*hours
Arm/Group | Arm A (Active-active) | Arm B (Placebo-active)
Number analyzed (Participants) | 47 | 47
Sum of scores*hours | 39.51 (55.416) | 47.21 (69.443)
Statistical Analysis 1: Comparison: Arm A (Active-active) vs Arm B (Placebo-active); Test type: Superiority; p = 0.729, ANCOVA; Least Square Mean Difference = -4.06, 95% CI 2-sided [-27.24 to 19.12], Standard Error of Mean 11.672 — Least-squares means, standard errors and p-value are taken from an analysis of covariance, with treatment group as fixed categorical effect and baseline TOSS (H0 at Day 1) as covariate

7. Secondary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any symptom, sign, illness or experience that develops or worsens in severity during the course of the study. A treatment emergent adverse event (TEAE) is an event that emerges during treatment, having been absent pretreatment, or worsens relative to the pretreatment state.
Time Frame: From Day 2 to Day 5
Population: The SAF set contained all participants in the ITT set who received at least one dose of study drug and participants were classified according to treatment received.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A (Active-active) | Arm B (Placebo-active)
Number analyzed (Participants) | 47 | 47
percentage of participants | 19.1 | 12.8

ADVERSE EVENTS:
Time Frame: From Day 2 to Day 5
Description: All-Cause Mortality, Serious Adverse Events and Other (Not Including Serious) Adverse Events is mentioned for Safety Analysis (SAF) Set. The SAF set contained all participants in the ITT set who received at least one dose of study drug and participants were classified according to treatment received.
Arm/Group | Arm A (Active-active) | Arm B (Placebo-active)
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/47
Other Adverse Events (participants affected / at risk) | 9/47 | 6/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Active-active) (N=47) | Arm B (Placebo-active) (N=47)
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Oedema mucosal (General disorders) | 2 | 0
Seasonal allergy (Immune system disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 2
Sinus headache (Nervous system disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2022-09-21): https://cdn.clinicaltrials.gov/large-docs/54/NCT05692154/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-17): https://cdn.clinicaltrials.gov/large-docs/54/NCT05692154/SAP_001.pdf